CLINICAL TRIAL: NCT01908790
Title: Correlation of Venous Oxygen Saturation Measurements by Non-invasive Mespere Venous Oximeter vs Venous Oxygen Saturation From Blood Samples From the Jugular Vein vs Central Venous Oxygen Saturation vs Mixed Venous Oxygen Saturation, Measured by a CO-Oximeter.
Brief Title: Correlation of Venous Oxygen Saturation Measurements by Non-invasive Mespere Venous Oximeter and Central Venous Catheter
Status: Completed | Type: Observational
Sponsor: Mespere Lifesciences Inc. (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Other Study IDs: HUM00075160
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Validation of Oximeter System
Keywords: venous oximeter; non-invasive monitor; heart failure (HF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heart Failure Patients: Acute and chronic heart failure patients already receiving right heart catheterization (RHC) as part of their usual care
  Interventions: Device: Mespere Venous Oximeter; Device: Avoximeter 4000

INTERVENTIONS:
Device: Mespere Venous Oximeter — The Mespere VA Oximeter System is a non-invasive medical device for measurement of venous blood oxygenation.
Device: Avoximeter 4000 — The portable Avoximeter 4000 provides rapid, accurate assessment of the patient's true oxygenation status at the bedside. Features: Results in less than 10 seconds; No sample preparation required; Uses whole blood sample; Easy to use.

SUMMARY:
The purpose of this study is to establish the accuracy of the non-invasive Mespere Oximeter that estimates venous oxygen saturation.

DETAILED DESCRIPTION:
The conventional pulse oximeter has been a standard in clinical care for non-invasive hemodynamic monitoring, which only measures arterial blood oxygenation. The clinical application of venous oximetry is numerous, including severe sepsis and septic shock, severe trauma and hemorrhagic shock, and heart failure and cardiac arrest.

The existing method for venous blood oxygenation monitored is either through an invasive fiber optic catheter, or intermittently by blood sampling and CO-Oximetry. However, catheterization can be costly and can include inherent risks. Therefore, due to the inherent risks of catheterization, venous oximetry is limited only to critically ill patients.

By non-invasively monitoring venous blood oxygenation, the Mespere Oximeter provides more complete information on patient hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Heart failure patients already receiving RHC as part of their usual care
* Signed written and informed consent

Exclusion Criteria:

* Lack of patient consent
* Subject is pregnant
* Evidence of abnormal neck anatomy
* Subject does not have visible left and right jugular veins
* Subject has occluded internal jugular veins under ultrasound imaging
* Allergic to adhesive tape
* Ongoing photodynamic therapy
* Presence of known anatomical shunt or AV dialysis fistula
* Known central vein stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute and chronic heart failure patients already receiving right heart catheterization (RHC) as part of their usual care
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Mespere Oximeter venous oxygen saturation accuracy compared to CO-Oximeter | 0-10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Todd M Koelling, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Cardiovascular Center, Ann Arbor, Michigan, United States